CLINICAL TRIAL: NCT05949229
Title: The Effect of Preoperative Duloxetine on the Occurance of Postoperative Delirium in Patients Undergoing Cancer Surgery .
Brief Title: The Effect of Preoperative Duloxetine on the Occurance of Postoperative Delirium in Patients Undergoing Cancer Surgery.
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amira Hassan Ahmed Ali (Other)
Responsible Party: Sponsor-Investigator, Amira Hassan Ahmed Ali, Egypt , Assiut governorate., Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pain management
Record Dates: First submitted 2023-07-10; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Post Operative Delirium
Keywords: Duloxetine, POD, postoperative dilrium
MeSH Terms: conditions — Emergence Delirium | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Intervention Model Description: The participating patients will be randomly allocated using computer generated randomizer program (http://www.randomizer.org) into 2 study groups . Duloxetine group (Group D): patients received oral duloxetine 60 mg 2 hours just before operation. Control group (Group C): patients received an identical placebo pill 2 hours just before operation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participating patients will be randomly allocated using computer generated randomizer program (http://www.randomizer.org) into 2 study groups .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Duloxetine group (Group D) (Experimental): patients received oral duloxetine 60 mg 2 hours just before operation.
  Interventions: Drug: Duloxetine 60 MG
- Control group (Group C) (Placebo Comparator): patients received an identical placebo pill 2 hours just before operation.
  Interventions: Drug: Duloxetine 60 MG

INTERVENTIONS:
Drug: Duloxetine 60 MG — Patients will recieve 2-hour preoperative duloxetine

SUMMARY:
This is prospective double-blinded placebo-randomized controlled trial that aims to compare the effect of preoperative administration of oral duloxetine 60 mg on decreasing the incidence of postoperative delirium in cancer patients undergoing surgery.

DETAILED DESCRIPTION:
This is prospective double-blinded placebo-randomized controlled trial that aims to compare the effect of preoperative administration of oral duloxetine 60 mg on decreasing the incidence of postoperative delirium in cancer patients undergoing surgery.

The participating patients will be randomly allocated using computer generated randomizer program (http://www.randomizer.org) into 2 study groups . Duloxetine group (Group D): patients received oral duloxetine 60 mg 2 hours just before operation. Control group (Group C): patients received an identical placebo pill 2 hours just before operation

Interventions:

The preoperative anaesthetic assessment will be carried out including patient medical history , examination including baseline heart rate and blood pressure recording and review of patients' CBC , coagulation profile and chemistry investagations. In the operating room in all patients a large bore IV access (18 gauge) will be inserted.

All patients will be connected to standard routine monitoring ( non-invasive blood pressure , electrocardiography and peripheral oxygen saturation) . patients will undergo surgery under general anasthesia [ induction with IV anaesthetics (propofol 2mg/kg ) , atracurium 0.5mg/kg and maintenance with inhalational anesthesia (sevoflurane and isoflurane ). patients will be transferred to ICU after surgery . CAM-ICU will be measured every eight hours (three times a day) until the patient wiil be discharged from the ICU. Positive CAM-ICU will be considered to be delirium.

Data collection:

Pre-operative data included: age, sex, ASA classification, smoking, tumor location , tumor stage, and history of medical disease. Intra-operative data included: duration of operation, blood loss, blood and fluid transfusion. Post-operative data included: length of hospital stay, and condition on discharge (living/dead).

Sample size:

Based on determining the main outcome variable, the estimated minimum required sample size is 42 patients (21 in each group).

The sample size was calculated using G*power software 3.1.9.2., based on the following assumptions:

Main outcome variable is the variation in CAM-ICU score used to evaluate postoperative delirium in cancer surgery patients who were administered preoperative duloxetine compared to those who received a placebo. Although no prior research has examined the impact of duloxetine on delirium, one study indicated that its use resulted in a considerably better postoperative recovery outcome than that of a placebo.(Hetta et al., 2020) Main statistical test is one-sided t-test to detect the difference between the two groups, Alpha = 0.05, Power = 0.80, Effect size = 0.8, Allocation ratio= 1

Statical analysis:

Data will be analyzed using IBT SPSS advanced statistics version200(spss inc,Chicago , il) . Numerical data will be expressed as mean and standard deviation or median and range as appropriate. Qualitative data will be expressed as frequency and percentage chi-square test(fisher's exact test) will be used to examine. The relation between qualitative variables for quantitative data, comparison between two groups will be done using independent sample test or Mann Whiteny test . a P value 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* All patients will sign an informed consent prior to inclusion in the study.
* Adult patients with ASA class I-III, undergoing cancer surgery.

Exclusion Criteria:

* Patients with pre-existing neuro- cognitive dysfunction.
* Documented signs of dementia after psychiatric evaluations.
* Language barriers or deafness.
* Psychosis stroke, meningitis, or brain tumors

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
postoperative delirium | 48 postoperative
  Patients that will recieve preoperative duloxetine will transported to ICU .CAM-ICU will be measured every eight hours (three times a day) until the patient wiil be discharged from the ICU. Positive CAM-ICU will be considered to be delirium.

CONTACTS AND LOCATIONS:
Overall Officials: Amira Hassan Ahmed, resident, Principal Investigator — Faculty of medecine,assiut,Egypt
Locations (1):
- Faculty of medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rodrigues-Amorim D, Olivares JM, Spuch C, Rivera-Baltanas T. A Systematic Review of Efficacy, Safety, and Tolerability of Duloxetine. Front Psychiatry. 2020 Oct 23;11:554899. doi: 10.3389/fpsyt.2020.554899. eCollection 2020. PMID 33192668
- [Result] Chen H, Jiang H, Chen B, Fan L, Shi W, Jin Y, Ren X, Lang L, Zhu F. The Incidence and Predictors of Postoperative Delirium After Brain Tumor Resection in Adults: A Cross-Sectional Survey. World Neurosurg. 2020 Aug;140:e129-e139. doi: 10.1016/j.wneu.2020.04.195. Epub 2020 May 4. PMID 32376378
- [Result] Dos Santos FCM, Rego AS, Montenegro WS, de Carvalho STRF, Cutrim RC, Junior AAM, Pereira FHF, Dibai-Filho AV, Bassi-Dibai D. Delirium in the intensive care unit: identifying difficulties in applying the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU). BMC Nurs. 2022 Nov 23;21(1):323. doi: 10.1186/s12912-022-01103-w. PMID 36419158
- [Result] Hetta DF, Elgalaly NA, Hetta HF, Fattah Mohammad MA. Preoperative Duloxetine to improve acute pain and quality of recovery in patients undergoing modified radical mastectomy: A dose-ranging randomized controlled trial. J Clin Anesth. 2020 Dec;67:110007. doi: 10.1016/j.jclinane.2020.110007. Epub 2020 Aug 22. PMID 32847776
- [Result] Ormseth CH, LaHue SC, Oldham MA, Josephson SA, Whitaker E, Douglas VC. Predisposing and Precipitating Factors Associated With Delirium: A Systematic Review. JAMA Netw Open. 2023 Jan 3;6(1):e2249950. doi: 10.1001/jamanetworkopen.2022.49950. PMID 36607634